CLINICAL TRIAL: NCT03090308
Title: Impact of Pulmonary Contusion in Patient's Outcome When Associated With Traumatic Flail Chest: An Observational Study
Brief Title: Pulmonary Contusion Flail Chest Complex
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Assistant professor of anesthesia and ICU, Assiut University
Other Study IDs: IRB0000871241
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Contusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Noninvasive positive pressure ventilation — All patients were ventilated using NIPPV (Engstrom Carestation), which was delivered to the patient through full-face mask and was started with pressure support of 8-12 cmH2O and PEEP of 3-5 cmH2O and gradually increased in 2 cmH2O steps. When patients tolerate FiO2 ≤ 0.5 with pressure support ≤ 8 cmH2O and PEEP ≤ 5 cmH2O for > 6 consecutive hours, withdrawal from NIPPV was attempted daily in 30 minutes spontaneous breathing trials.

SUMMARY:
The study included 20 adult patients presented by multiple fractured ribs (flail segment) with thoracic trauma severity score (TTSS) between 5 and 15. All patients received mid-thoracic epidural analgesia with 0.125% Bupivacaine and 1 μg/ml fentanyl. The patients were ventilated using non-invasive positive pressure ventilation (NIPPV). Follow up arterial blood gases, chest X-ray and CT scan were obtained. Parameters to be recorded: Patient's characteristics and clinical data including pulmonary contusion, number of fractured ribs, pleural involvement, PaO2/FiO2 ratio on admission, weaning outcome, duration of NIPPV, length of stay in ICU (LOS ICU), complications and mortality rate.

DETAILED DESCRIPTION:
20 Patients fulfilling the inclusion criteria were submitted to strapping and packing in the form of dressing and fixing with elastoplast. All patients were ventilated using NIPPV (Engstrom Carestation), which was delivered to the patient through full-face mask and was started with pressure support of 8-12 cmH2O and PEEP of 3-5 cmH2O and gradually increased in 2 cmH2O steps. When patients tolerate FiO2 ≤ 0.5 with pressure support ≤ 8 cmH2O and PEEP ≤ 5 cmH2O for > 6 consecutive hours, withdrawal from NIPPV was attempted daily in 30 minutes spontaneous breathing trials. Therapy was considered successful if endotracheal intubation was avoided and the patient could be discharged from the ICU. During this period follow up arterial blood gases, chest X-rays and CT scans were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple fractured ribs with flail segment presented by acute respiratory distress that had deteriorated despite effective pain management, their age more than 18 years and less than 70 years, with thoracic trauma severity score (TTSS) between 5 and 15

Exclusion Criteria:

* Patients requiring endotracheal intubation or emergency surgery following admission, severe associated trauma to other systems, respiratory failure caused by neurological disease or asthmatic attack or any contraindication for NIPPV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 Patients fulfilling the inclusion criteria were submitted to strapping and packing in the form of dressing and fixing with elastoplast. All patients were ventilated using NIPPV (Engstrom Carestation), which was delivered to the patient through full-face mask and was started with pressure support of 8-12 cmH2O and PEEP of 3-5 cmH2O and gradually increased in 2 cmH2O steps. When patients tolerate FiO2 ≤ 0.5 with pressure support ≤ 8 cmH2O and PEEP ≤ 5 cmH2O for > 6 consecutive hours, withdrawal from NIPPV was attempted daily in 30 minutes spontaneous breathing trials. Therapy was considered successful if endotracheal intubation was avoided and the patient could be discharged from the ICU. During this period follow up arterial blood gases, chest X-rays and CT scans were obtained.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
PaO2 mmHg | 24 hours after starting NIPPV
  The correlations of pulmonary contusion with PaO2

SECONDARY OUTCOMES:
PaO2/FiO2 ratio | 24 hours after starting NIPPV
  The correlations of pulmonary contusion with PaO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Abdelraheem, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301